CLINICAL TRIAL: NCT01602744
Title: The Use of STOPP/START Criteria for Medication Intervention and the Risk of Falls, Hospitalization, Functioning and Quality of Life Among Elderly Population Living in a Geriatric Hospital in Israel and Comparison to Beers
Brief Title: The Use of STOPP/START Criteria for Medication Intervention Among Elderly Population Living in a Geriatric Hospital
Acronym: STOPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 0036-12 WOMC
Record Dates: First submitted 2012-05-01; First posted 2012-05-21 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Adverse Drug Effects
Keywords: STOPP screening tool; START screening tool; MIP-medication inappropriate prescription; PIM-Potentially inappropriate medication
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Potentially Inappropriate Medication List

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controll (No Intervention): The medications in this arm will not be screened.
- Intervention screening medication group (Active Comparator): STOPP/START screening tools are used for medication intervention
  Interventions: Other: STOPP/START screening tools for medication intervention

INTERVENTIONS:
Other: STOPP/START screening tools for medication intervention — In the intervention arm the investigator will use the screening tools STOPP/START to screen the medications.
  Other Names: STOPP Criteria; START Criteria; medication intervention
  Arms: Intervention screening medication group

SUMMARY:
The purpose of this study is to determine if the use of STOPP/START criteria (STOPP-screening tool of older persons potentially inappropriate prescriptions START-screening tool to alert doctors to right treatment)for medication intervention in elderly population living in a geriatric hospital will lower the number of falls,hospitalization,will improve functioning, quality of life and reduce financial costs.

DETAILED DESCRIPTION:
Inappropriate prescribing is common in older people and is associated with adverse drug effects,hospitalization and falls. In this trial we want to check the efficacy of the screening tools STOPP/START which were developed and validated in order to reduce inappropriate prescribing. STOPP comprises of 65 indicators of drug-drug, drug-disease interactions and therapeutic duplication. START incorporates 22 evidence based indicators of common prescribing omissions. We will conduct a randomized controlled trial to test the hypothesis that screening the medications of older patients living permanently in a geriatric hospital will improve their quality of life. The compliance of the doctor working in the geriatric hospital to the recommendations of the screening tools will also be checked.

ELIGIBILITY:
Inclusion Criteria:

* age over 65
* live in the geriatric hospital "Givaat Hashlosha" permanently.

Exclusion Criteria:

* people with a terminal illness that will not live more than a year.
* people who enter the geriatric hospital for a short while (are not permanent).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 382 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariella Herskowits, MBA, Principal Investigator — Wolfson Medical Center
Locations (1):
- Givaat Hashlosha Geriatric Hospital, Petah Tikva, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected on April 2012 from 382 residents' records in "Givaat Hashlosha" geriatric facility.23 residents were excluded for not fulfilling study entry criteria. The final study group was comprised of 359 residents. 359 residents were randomized on May 2012 to recieve either STOPP/START screening (N=183) or usual care (n=176).
Pre-assignment Details: 23 residents were excluded: 10 were younger than 65 years of age, one was not taking medications, 5 had a terminal illness and 7 had been on a short stay in the facility.
Groups:
- Intervention STOPP/START: Screening medications with STOPP/START critera
Period: Overall Study
Arm/Group | Controll | Intervention STOPP/START
Started | 176 | 183
Completed | 146 | 160
Not Completed | 30 | 23
Not completed — Death | 17 | 15
Not completed — Lost to Follow-up | 13 | 8

BASELINE CHARACTERISTICS:
Population: All residents in the geriatric facility (382) were recruited for the trial. 23 were excluded for not fulfilling study entry criteria. The final study group was comprised of 359 residents. Residents were randomized to recieve either STOPP/START screening (intervention, n=183) or usual care (control, n=176).
Groups:
- Total: Total of all reporting groups
Arm/Group | Controll | Intervention STOPP/START | Total
Number analyzed (Participants) | 176 | 183 | 359
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 176 | 183 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.2 (9.4) | 83.1 (7.99) | 82.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 129 | 239
  Male | 66 | 54 | 120
Region of Enrollment [Number; unit: participants]
  Israel | 176 | 183 | 359

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life- Mental Component Summaty (MCS)
Description: Quality of life will be measured by MOS SF-12 Health Survey questionnare. Results are expressed in terms of two meta scores: The Physical Component Summary(PCS) and the Mental Component Summary (MCS). The PCS and MCS scores have a range of 0 to 100, thus scores greater than 50 represent a better than average health status.
Time Frame: Outcome measures were assessed at the end of the 12 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controll | Intervention STOPP/START
Number analyzed (Participants) | 146 | 160
units on a scale | 39.6 (11.3) | 37.7 (11.69)

2. Secondary Outcome: Pharmacoeconomics Analysis-Costs of Medication
Description: The costs on medications in the geriatric hospital before and after intervention e.g. pharmaeconomic analysis of the intervention. Costs of medications were calculated in New Israeli shekels per month and taken from the Ministry of Health's medication price list.
Time Frame: Outcome measures were assessed at the end of the 12 month follow up
Measure: Mean (Standard Deviation); unit: New Israeli shekels per month
Arm/Group | Controll | Intervention STOPP/START
Number analyzed (Participants) | 146 | 160
New Israeli shekels per month | 402.3 (291.2) | 279 (171.9)

3. Primary Outcome: SF-12 Health Survey questionnaire-the Physical Component Summary (PCS)
Description: Quality of life was assessed by the SF-12 Health Survey questionnare. Results are expressed in terms of two meta scores:the Physical Component Summary (PCS) AND Mental Component Summary (MCS). The PCS and MCS scores have a range of 0 to 100, thus scores greater than 50 represent a better than average health status.
Time Frame: Outcome measures were assessed at the end of the 12 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controll | Intervention STOPP/START
Number analyzed (Participants) | 146 | 160
units on a scale | 33 (8.3) | 33.1 (8.1)

4. Primary Outcome: Falls
Description: Average number of falls per year.
Time Frame: At the end of the 12 month follow up
Measure: Mean (Standard Deviation); unit: Number of falls per year
Arm/Group | Controll | Intervention STOPP/START
Number analyzed (Participants) | 146 | 160
Number of falls per year | 1.26 (2.4) | 0.8 (1.34)

5. Primary Outcome: Hospitalizations
Description: The average number of hospitalizations per year.
Time Frame: Outcome measures were assessed at the end of the 12 month follow up
Measure: Mean (Standard Deviation); unit: Number of hospitalizations per year
Arm/Group | Controll | Intervention STOPP/START
Number analyzed (Participants) | 146 | 160
Number of hospitalizations per year | 0.47 (0.87) | 0.49 (1.05)

6. Primary Outcome: Functional Independence Measure (FIM)
Description: Functioning was assessed by the FIM score. The FIM rates 18 activities of daily living on a 7 point scale ranging from fully dependent (=1) to independent (=7). A maximum score of 126 indicates functional independence and the lowest score of 18 indicates functional dependence.
Time Frame: Outcome measures were assessed at the end of the 12 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controll | Intervention STOPP/START
Number analyzed (Participants) | 146 | 160
units on a scale | 55.4 (36.8) | 54.3 (35.1)

ADVERSE EVENTS:
Time Frame: One year of follow up.
Description: A daily follow up of the chief physician un the geriatric facility.
Arm/Group | Controll | Intervention STOPP/START
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/183
Other Adverse Events (participants affected / at risk) | 0/176 | 0/183

LIMITATIONS AND CAVEATS:
The limitations of the study were that it was conducted in a single geriatric center. This precludes the possibility of generalizing its findings to other older segments of the community.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No